CLINICAL TRIAL: NCT00571766
Title: Effects of Oral L-Arginine on Chronic Hypertension in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Fabio Facchinetti, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oral L-Arginine
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension in Pregnancy
Keywords: chronic hypertension in pregnancy; chronic Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral L-Arginine 2 g twice a day for 14 weeks
  Interventions: Drug: L-Arginine
- 2 (Placebo Comparator): Placebo 2 g, twice a day for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Arginine — Oral L-Arginine 2g, twice a day for 14 weeks
  Arms: 1
Drug: Placebo — Placebo 2 g twice a day for 14 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effects of oral L-Arginine in pregnant women with chronic hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18-20 week of gestation with chronic hypertension

Exclusion Criteria:

* Maternal or fetal disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to evaluate blood pressure changes in pregnant women with chronic hypertension during oral arginine or placebo treatment in second trimester of gestation. | 14 weeks

SECONDARY OUTCOMES:
To evaluate if is necessary add a conventional therapy for hypertension, to evaluate the maternal and fetal outcomes and possible complications, to evaluate the safety of L-Arginine. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Facchinetti, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- University of Modena and Reggio Emilia, Modena, Emilia-Romagna, Italy